CLINICAL TRIAL: NCT00456053
Title: A Randomized Study of the Safety and Efficacy of FG-2216 in Subjects With Renal Anemia Not Requiring Dialysis and Not Receiving Recombinant Human Erythropoietin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: FGCL-SM2216-019
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Renal Anemia
Keywords: Renal Anemia; Renal Failure; Kidney Disease; Human EPO
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: FG2216

SUMMARY:
The purpose of this study is to test the safety and efficacy of FG-2216 in the treatment of patients with renal anemia who are not receiving erythropoietin and who are not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 or 4 chronic kidney disease
* appropriate hemoglobin levels

Exclusion Criteria:

* Neovascular age related macular degeneration requiring treatment
* Macular edema or proliferative retinopathy in diabetic subjects, requiring treatment
* Any history of malignancy
* Therapy with recombinant erythropoietin or red blood cell transfusion within 4 weeks
* Renal Transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2005-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (Hb) response

SECONDARY OUTCOMES:
Attainment of Hb target range (11-13)
Duration of maintenance of Hb in target range (11-13)
Safety

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - 3 Research Sites, Los Angeles, California
  - Research Site, Oakland, California
  - Research Site, San Diego, California
  - Research Site, Santa Clara, California
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, South Holland, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Springfield, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Flushing, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Fairfax, Virginia